CLINICAL TRIAL: NCT06222489
Title: Whole Body HER3 Quantification With Radiolabelled Patritumab Deruxtecan (HER3-DXd) PET/CT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N23HDX
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Carcinoma; Advanced Non-Small Cell Squamous Lung Cancer; EGFR Gene Mutation
Keywords: At least one line of systemic treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Product Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patritumab Deruxtecan (Other): 5.6 mg/kg patritumab deruxtecan every 3 weeks
  Interventions: Drug: 89Zr-Patritumab deruxtecan

INTERVENTIONS:
Drug: 89Zr-Patritumab deruxtecan — Day 1, day 3, day 6, day 11 and day 26 of first course
  Other Names: Tracer

SUMMARY:
Activity of patritumab deruxtecan (U3-1402; HER3-DXd) has been shown in a phase I/II study in patients with HER3 expressing breast cancer as well as in a phase I study in patients with EGFR TKI refractory EGFR mutation positive NSCLC with a preliminary ORR of 25%. HER3 expression can be seen in multiple tumor types and is therefore an attractive target for antibody drug conjugate (ADC) treatment. However, intra- and intertumor heterogeneity of HER3 expression might be substantial, as is seen for HER2, and might contribute to treatment failure or heterogeneous responses. In addition, HER3 expression is dynamic and has been shown to change over time.

In order to identify patients that may benefit most from treatment with patritumab deruxtecan, better knowledge of the in vivo behaviour of the drug is warranted. One way to visualize this behaviour is positron emission tomography (PET) imaging with radiolabelled antibodies (immune-PET). 89Zr-Patritumab deruxtecan PET/CT can assess HER3 expression non-invasively at a whole body level, including sites that may be difficult to biopsy. It also visualizes and quantifies biodistribution of patritumab deruxtecan, thereby obtaining valuable information for safety and toxicity analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Have a histologically or cytologically confirmed diagnosis of (locally) advanced stage EGFR mutation positive NSCLC, not amenable for curative intent treatment.
3. Have measurable disease according to RECIST 1.1.
4. At least two lesions with a long axis diameter ≥2 cm.
5. Have received at least one line of EGFR TKI treatment for (locally) advanced stage NSCLC.
6. In case the tumor is positive for T790M mutation, prior treatment with a third generation EGFR TKI is mandatory.
7. Patients must be ≥18 years of age.
8. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1 at the time of Screening.
9. Has adequate bone marrow reserve and organ function, based on local laboratory data within 14 days prior to Cycle 1, Day 1, defined as:

   * Platelet count ≥100 000/mm3 or ≥100 × 109/L (platelet transfusions are not allowed up to 14 days prior to Cycle 1 Day 1 to meet eligibility)
   * Hemoglobin (Hgb) ≥9.0 g/dL or 5.6 mmol/L (transfusion and/or growth factor support is allowed)
   * Absolute neutrophil count (ANC) ≥1500/mm3 or ≥1.5 × 109/L
   * Creatinine clearance (CrCl) ≥30 mL/min as calculated using the Cockcroft-Gault equation or measured CrCl
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤3 × ULN (if liver metastases are present, ≤5 ×ULN)
   * Total bilirubin (TBL) ≤1.5 × ULN if no liver metastases (<3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases)
   * Serum albumin ≥2.5 g/dL or 25 g/L
   * Prothrombin time (PT) or Prothrombin time- international normalized ratio (PT-INR) and activated partial thromboplastin time (aPTT)/partial thromboplastin time (PTT) ≤1.5 × (ULN), except for subjects on coumarin-derivative anticoagulants or other similar anticoagulant therapy, who must have PT-INR within therapeutic range as deemed appropriate by the Investigator
10. Be willing to provide a qualifying tumor tissue specimen. A pretreatment tumor biopsy (if medically feasible) or otherwise archival tumor tissue is required. Samples must be of sufficient quantity and of adequate tumor tissue content (as defined in the Laboratory Manual).

    1. A Baseline pretreatment tumor biopsy must be of the primary (if intact) and/or metastatic lesion(s) not previously irradiated and amenable to core biopsy. Any serious adverse event (SAE) directly related to the new biopsy should be reported as outlined in Section 8.
    2. If not medically feasible to collect the pretreatment tumor biopsy, archival tumor tissue not previously irradiated must be collected from a biopsy on or after treatment with the most recent EGFR TKI cancer therapy regimen.
11. If the subject is a female of childbearing potential, she must have a negative serum pregnancy test at screening and must be willing to use a highly effective birth control upon enrollment, during the Treatment Period, and for 7 months, following the last dose of study drug. A female is considered of childbearing potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months) unless permanently sterile (undergone a hysterectomy, bilateral salpingectomy or bilateral oophorectomy) with surgery at least 1 month before the first dose or confirmed by follicle stimulating hormone (FSH) test.
12. Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration.
13. If male, the subject must be surgically sterile or willing to use a highly effective birth control upon enrollment, during the treatment period, and for at least 4 months following the last dose of study drug.
14. Male subjects must not freeze or donate sperm starting at screening and throughout the study period, and for at least 4 months after the final study drug administration.

Exclusion Criteria:

1. Any history of interstitial lung disease (ILD) (including pulmonary fibrosis or radiation pneumonitis), has current ILD, or is suspected to have such disease by imaging during screening.
2. Clinically severe pulmonary compromise (based on investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

   1. any underlying pulmonary disorder (eg, pulmonary emboli, severe asthma, severe chronic obstructive lung disease (COPD), restrictive lung disease, pleural effusion);
   2. any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement (eg, rheumatoid arthritis, Sjögren's syndrome, sarcoidosis); OR prior pneumonectomy.
3. Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent or any form of immunosuppressive therapy prior to Cycle 1 Day 1. Subjects who require use of bronchodilators, inhaled steroids, or local steroid injections may be included in the study.
4. Evidence of any leptomeningeal disease.
5. Has clinically significant corneal disease.
6. Any evidence of severe or uncontrolled systemic diseases (including active bleeding diatheses, active infection, psychiatric illness/social situations, geographical factors, substance abuse, or other factors which in the Investigator's opinion makes it undesirable for the subject to participate in the study or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required.
7. Evidence of clinically active spinal cord compression or brain metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Subjects with clinically inactive or treated brain metastases who are asymptomatic (ie, without neurologic signs or symptoms and do not require treatment with corticosteroids or anticonvulsants) may be included in the study. Subjects must have a stable neurologic status for at least 2 weeks prior to Cycle 1 Day 1.
8. Inadequate washout period prior to Cycle 1 Day 1, defined as:

   1. Whole brain radiation therapy <14 days or stereotactic brain radiation therapy <7 days.
   2. Any cytotoxic chemotherapy, investigational agents or other anticancer drug(s) from a previous cancer treatment regimen or clinical study (other than Epidermal growth factor receptor tyrosine kinase inhibitor (EGFR TKI)), <14 days or 5 half-lives, whichever is longer.
   3. Monoclonal antibodies other than immune checkpoint inhibitors, such as bevacizumab (anti-VEGF) and cetuximab (anti-EGFR) <28 days.
   4. Immune checkpoint inhibitor therapy < 21 days.
   5. Major surgery (excluding placement of vascular access) < 28 days.
   6. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation < 28 days or palliative radiation therapy < 14 days.
   7. Chloroquine or hydroxychloroquine ≤ 14 days.
9. Prior treatment with an HER3 antibody and/or antibody drug conjugate (ADC) that consists of an exatecan derivative that is a topoisomerase I inhibitor (eg, trastuzumab deruxtecan).
10. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, grade ≤1 or baseline. Subjects with chronic Grade 2 toxicities may be enrolled at the discretion of the Investigator after consultation with the Sponsor Medical Monitor or designee.
11. Has known hypersensitivity to either the drug substances or inactive ingredients in the drug product.
12. Has any primary malignancy other than locally advanced or metastatic NSCLC within 3 years prior to Cycle 1 Day 1, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated.
13. Uncontrolled or significant cardiovascular disease prior to Cycle 1 Day 1, including:

    1. QT interval corrected by Fridericia's formula (QTcF) prolongation interval of >470 ms for females and >450 ms for males.
    2. Left ventricular ejection fraction (LVEF) <50% by either echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan.
    3. Resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg.
    4. Myocardial infarction within 6 months.
    5. New York Heart Association (NYHA) Classes 2 to 4 within 28 days.
    6. Uncontrolled angina pectoris within 6 months.
    7. Cardiac arrhythmia requiring antiarrhythmic treatment.
14. Active Hepatitis B and/or Hepatitis C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1, Day 1.

    a. Subjects with past or resolved Hepatitis B virus (HBV) infection are eligible if: i. Hepatitis surface antigen (HBsAg) negative and hepatitis B core antibody (anti-HBc) positive; OR ii. HBsAg positive and HBV DNA viral load is documented to be ≤ 2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with normal transaminases (in the absence of liver metastasis); OR iii. HBsAg positive and HBV DNA viral load is documented to be ≤ 2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with liver metastasis and abnormal transaminases AST/ALT < 3 ULN.

    b. Subjects with a history of Hepatitis C infection will be eligible for enrollment only if the viral load according to local standards of detection, is documented to be below the level of detection in the absence of anti-viral therapy during the previous 12 weeks (ie, sustained viral response according to the local product label but no less than 12 weeks, whichever is longer).
15. Female subject who is pregnant or breastfeeding or intends to become pregnant during the study.
16. Subjects with known human immunodeficiency virus (HIV) infection.
17. Prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's judgment, could affect the safety of the subject; alter the absorption, distribution, metabolism or excretion of the study drug; or confound the assessment of study results.
18. Live virus vaccination 28 days prior to Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
The optimal imaging dose patritumab deruxtecan to co-inject with 89Zr-Patritumab deruxtecan (HER3-DXd), defined by adequate visualisation of the circulation five days after tracer injection. | From the date of cycle 1, day 1 until the date of cycle 1, day 5.
  Identification of the optimal non-radiolabeled patritumab deruxtecan dose to be co-injected with 89Zr-Patritumab deruxtecan to allow optimal 89Zr-Patritumab deruxtecan PET imaging.

SECONDARY OUTCOMES:
SUV of tumor lesions | From the date of cycle 1, dag 3 or 6 and cycle 1, day 14 or 17 and cycle 1, day 29 or 32.
  Quantify tumor 89Zr-Patritumab deruxtecan uptake (visually and quantitatively, expressed as SUV).

CONTACTS AND LOCATIONS:
Overall Officials: Joop de Langen, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
To be decided